CLINICAL TRIAL: NCT04573049
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Effectiveness and Safety of Levosimendan in Patients With Severe Aortic Stenosis and Heart Failure Undergoing Transcatheter Aortic Valve Replacement
Brief Title: The Effectiveness and Safety of Levosimendan in Patients With Severe Aortic Stenosis and Heart Failure Undergoing Transcatheter Aortic Valve Replacement
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: China International Medical Foundation (Other)
Responsible Party: Principal Investigator, Jianhui Wang, Principle Investigator and Clinical professor, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020-1357
Record Dates: First submitted 2020-09-15; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Aortic Valve Stenosis; Heart Failure; Inotropic Agents; Safety Issues; Effect of Drug; Cardiac Event; Transcatheter Aortic Valve Replacement
Keywords: Aortic valve stenosis; Heart failure; Levosimendan; Transcatheter Aortic Valve Replacement; Effectiveness; Safety; NT-proBNP
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Failure; Cardiovascular Diseases | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levosimendan (Experimental): Levosimendan 0.1µg/kg/min will last for 24h after the valve is released.
  Interventions: Drug: Levosimendan
- Placebo (Placebo Comparator): 5% glucose 0.1µg/kg/min administration will continue for 24h after the valve is released.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Levosimendan — On the basis of routine care given by corresponding clinicians, 0.1µg/kg/min levosimendan is given for 24 hours.
  Arms: Levosimendan
Other: Placebo — On the basis of routine care given by corresponding clinicians, 0.1µg/kg/min 5% glucose infusion is given for 24 hours.
  Arms: Placebo

SUMMARY:
A study to evaluate the effectiveness and safety of levosimendan compared with placebo in subjects with severe aortic stenosis and heart failure undergoing transcatheter aortic valve replacement

DETAILED DESCRIPTION:
The number of subjects undergoing transcatheter aortic valve replacement to treat aortic stenosis have been increasing in recent decades. Levosimendan, an innovative inotrope, is powerfully evidenced to have the function to improve cardiac output and hemodynamic parameters. However, there is no specified study concentrated on the role of Levosimendan in surgical procedure such as transcathter aortic intervention. This double-blind, randomized, placebo-controlled study is aimed to investigate the effectiveness and safety of Levosimendan in adults having severe aortic stenosis combined with heart failure undergoing transcatheter aortic valve replacement. Therefore, the purpose of this trial is to explore whether the improvement of cardiac and renal performance can be rendered by intra-operative Levosimendan infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Signed (by the subjects or their legally acceptable representatives) informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study
2. Severe aortic stenosis

   1. Mean transaortic gradient ≥ 40 mmHg(at rest or stress)
   2. Aortic peak velocity ≥ 4m/s;
   3. Arotic valve area <0.8 cm2 and/or aortic valve area index< 0.5cm2/m2
3. Cardiac dysfunction

   1. LVEF≤50% (estimated by Simpson)
   2. NT-proBNP≥1500ng/L；
   3. Symptoms of dyspnea and fatigue when at rest or after slight exertion (New York Heart Association ≥ Ⅲ -Ⅳ)
   4. Intermittant fluid retention and/or symptoms induced by low cardiac output at rest, but lack of hemodynamic instability

Exclusion Criteria:

1. Decompensated acute cardiac failure due to hemodynamic instability
2. A historty of torsade de points ventricular tachycardia
3. Known allergic reaction or sensitivity to Levosimendan or excipients
4. Received levosimendan within 1 week prior to the planned clinical trial
5. Serum potassium < 3.5 mmol/L and > 5.5 mmol/L before the drug study
6. Systolic blood pressure < 90mmHg at baseline
7. Estimated glomerular filtration rate (eGFR) ≤30 mL/min/1.73m2.
8. Unable to participate in study for being critically ill asssed by clinicians
9. Other concomitant severe morbidities leading to poor prognosis and decreased mortality, such as malignant tumor and disease involving other vital organs; life expectancy less than 1 year.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
The change of NT-proBNP level | day 1, day 3, day 5, month 1 and month 3

SECONDARY OUTCOMES:
The change of CK-MB | day 1, day 3, day 5, month 1 and month 3
The change of c-TnI | day 1, day 3, day 5, month 1 and month 3
The change of left ventricular ejection fraction | day 1, day 3, day 5, month 1 and month 3
  It is evaluated by echcardiography.
The change of left ventricular end-diastolic diameter | day 1, day 3, day 5, month 1 and month 3
  It is evaluated by echcardiography.
The number of patients in need of secondary intra-operative vasoactive-inotropic substances | Peri-operation
  Vasoactive-inotropic substances include dobutamine, milrinone, epinephrine, dopamine and vasopressors.
The incidence of postoperative kidney injury | day 1, day 3, day 5, month 1 and month 3
  The kidney injury will be assessed by the change of serum creatinine, urea nitrogen and cystatin C.

OTHER OUTCOMES:
The incidence of adverse events | Peri-operation
  Adverse events include hypotension and arrythmia.
The incidence of atrial fibrillation | Peri-operation
The change of electrolyte | Peri-operation
  The change of electrolyte is evaluated by potassium, calcium and lactic acid level.
The number of patients having liver dysfunction | Peri-operation
  Liver dysfunction is assessed by the change of alanine aminotransferase (ALT) and aspartate aminotransferase (AST).
The length of intensive care unit stay | From date of surgery until intensive care unit discharge (assessed up to 1 month)
In-hospital medical expense | From baseline until hospital discharge (assessed up to 1 month)

CONTACTS AND LOCATIONS:
Locations (1):
- Jianhui Wang, Beijing, Beijing Municipality, China